CLINICAL TRIAL: NCT02816736
Title: EntrestoTM (LCZ696) In Advanced Heart Failure (LIFE Study)
Acronym: HFN-LIFE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00071722; 5U01HL084904 (NIH)
Record Dates: First submitted 2016-06-13; First posted 2016-06-29 (Estimated); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Heart Diseases; Cardiovascular Diseases; Valsartan; Entresto
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LCZ696 (Entresto) + placebo (Active Comparator): LCZ696 50 mg, 100 mg, or 200 mg orally twice daily for 24 weeks, plus valsartan placebo (to match 40 mg, 80 mg, or 160 mg) orally twice daily for 24 weeks
  Interventions: Drug: LCZ696; Drug: valsartan placebo
- valsartan + placebo (Active Comparator): valsartan 40 mg, 80 mg, or 160 mg orally twice daily for 24 weeks, plus LCZ696 placebo (to match 50 mg, 100 mg, or 200 mg) orally twice daily for 24 weeks
  Interventions: Drug: valsartan; Drug: LCZ696 placebo

INTERVENTIONS:
Drug: LCZ696 — Subjects previously taking no or low-dose ACEI or ARB, or who have an eGFR < 30 mL/min/1.73m²: starting dose of LCZ696 = 50 mg po BID.
  Subjects taking an ARB at greater than low dose: starting dose of LCZ696 = 100 mg po BID.
  Subjects taking an ACEI at greater than low dose: starting dose of LCZ696 = 100 mg po BID.
  * At Investigator discretion, study drug may be started at the low dose if there are any concerns regarding tolerability.
  Dose adjustments will be performed every 2 weeks by doubling the dose of LCZ696 up to the target max dose of 200 mg po BID as tolerated.
  The doses of LCZ696 are 50mg (one low-dose (50mg) tablet), 100mg (one high-dose (100mg) tablet), and 200mg (two high-dose (100mg) tablets.) These doses are equivalent to 24/26 mg, 49/51 mg, and 97/103 mg commercial Entresto™, respectively.
  Other Names: Entresto
  Arms: LCZ696 (Entresto) + placebo
Drug: valsartan — Subjects previously taking no or low-dose ACEI or ARB, or who have an eGFR < 30 mL/min/1.73m²: the starting dose of valsartan = 40 mg po BID.
  Subjects taking an ARB at greater than low dose: starting dose of valsartan = 80 mg po BID.
  Subjects taking an ACEI at greater than low dose: starting dose of valsartan = 80 mg po BID.
  * At Investigator discretion, study drug may be started at the low dose if there are any concerns regarding tolerability.
  Dose adjustments will be performed every 2 weeks by doubling the dose of valsartan up to the target maximum dose of 160 mg po BID, as tolerated.
  The doses of valsartan are 40mg (one low-dose (40mg) tablet), 80mg (one high-dose (80mg) tablet), and 160mg (two high-dose (80mg) tablets).
  Other Names: Diovan
  Arms: valsartan + placebo
Drug: LCZ696 placebo — LCZ696 placebo tablets will be supplied to match the low-dose (50mg) and high-dose (100mg) active LCZ696 tablets. Dosing for LCZ696 placebo will mirror dosing for active valsartan (the same number of low or high-dose tablets will be given.)
  Arms: valsartan + placebo
Drug: valsartan placebo — Valsartan placebo tablets will be supplied to match the low-dose (40mg) and high-dose (80mg) active valsartan tablets. Dosing for valsartan placebo will mirror dosing for active LCZ696 (the same number of low or high-dose tablets will be given.)
  Arms: LCZ696 (Entresto) + placebo

SUMMARY:
The primary objective of the study is to determine whether, in patients with symptomatic, advanced heart failure due to left ventricular systolic dysfunction, treatment with LCZ696 for 24 weeks will improve Pro-B-type Natriuretic Peptide (NT-proBNP) levels, which reflect hemodynamic and clinical status, compared to treatment with valsartan.

DETAILED DESCRIPTION:
Patients with advanced heart failure with reduced ejection fraction (HFrEF) have extremely high morbidity and mortality with 1 year outcomes of death and hospitalization of approximately 50%. For the most advanced heart failure patients, the evidence base for medical treatment is limited with consensus guidelines recommending consideration for either cardiac transplant or ventricular assist device, or palliative care.

The PARADIGM-HF trial showed that LCZ696, which consists of the neprilysin inhibitor sacubitril and the ARB valsartan, improved morbidity and mortality in patients with chronic HFrEF in comparison to enalapril. However, limited experience with advanced heart failure patients was gained from patients enrolled in the trial. Because the information on the effects of sacubitril/valsartan in patients with NYHA class IV heart failure is limited, the updated 2016 ACC/AHA/HFSA guidelines for the treatment of heart failure do not yet endorse the use of sacubitril/valsartan in patients with NYHA class IV heart failure. Accordingly, experience is needed on the use of, and outcomes with LCZ696 in patients unable to tolerate target doses of angiotensin-converting enzyme inhibitor (ACEI)/ angiotensin receptor blocker (ARB).

This study will be a randomized, double-blinded trial of advanced heart failure subjects with 1:1 randomization to either LCZ696 (sacubitril and valsartan) or valsartan. Study drug will be administered in a double-dummy fashion, in which subjects take active (LCZ696 or valsartan) and placebo. Approximately 400 subjects will be randomized into the study.

Subjects will have an initial screening evaluation, including baseline laboratory tests as well as an assessment of left ventricular (LV) ejection fraction, at which time preliminary subject eligibility will be determined. The LV ejection fraction may have been obtained within the prior 12 months by 2-D echocardiogram, LV angiogram or radionuclide scintigraphy. Willing subjects meeting entry criteria will be consented. Those who meet all entry criteria and are interested in study participation will be enrolled.

Enrolled subjects will complete baseline assessments and undergo a run-in period of 3-7 days with LCZ696 50 mg (equivalent to Entresto™ 24/26 mg) po BID (taken by mouth twice a day) prior to randomization. For subjects taking an ACEI, the ACEI will be withheld for ≥ 36 hours prior to first dose of LCZ696.

Subjects who tolerate the run-in period with LCZ696 will be randomized 1:1 to LCZ696 or valsartan.

Study treatment will be titrated to the target dose of 200 mg LCZ696 (equivalent to Entresto™ 97/103 mg) as two 100 mg LCZ696 and 2 placebo tablets po BID or valsartan 160 mg (two 80 mg valsartan and 2 placebo tablets) po BID.*

Randomized subjects will receive the first dose of study drug as follows:

* For subjects not previously taking ACEI or ARB, previously taking ACEI or ARB at a low dose*, or subjects who have an eGFR < 30 mL/min/1.73m², the starting dose of valsartan will be 40 mg po BID and the starting dose of LCZ696 will be 50 mg po BID.
* For subjects taking an ARB at greater than low dose†, the starting dose of valsartan will be 80 mg po BID and the starting dose of LCZ696 will be 100 mg po BID.*
* For subjects taking an ACEI at greater than low dose†, the ACEI will be withheld for ≥ 36 hours prior to randomization. The starting dose of valsartan will be 80 mg po BID and the starting dose of LCZ696 will be 100 mg po BID.*

  * At Investigator discretion, study drug may be started at the low dose (LCZ696/placebo 50 mg po BID or valsartan/placebo 40 mg po BID) if there are any concerns regarding tolerability at the 100 mg / 80 mg dose.)

Per package insert, the valsartan compounded in Entresto™ is more bioavailable than the valsartan in other marketed formulations. The dose equivalence for valsartan compounded in Entresto™ compared to valsartan prepared alone (Entresto™ dose = marketed valsartan dose) is as follows: 26 mg=40 mg, 51 mg=80 mg, 103 mg=160 mg.

† Low dose is defined as 24 hour dose of ≤ 10 mg lisinopril, ≤ 5 mg ramipril, ≤ 50 mg losartan, ≤ 10 mg olmesartan, or other dose equivalent.

Dose adjustments will be performed every 2 weeks by doubling the dose of LCZ696 or valsartan up to the target maximum dose. The doses of LCZ696 are 50 mg (one 50 mg active and 1 placebo tablet), 100 mg (one 100 mg active and 1 placebo tablet) and 200 mg (two 100 mg active and 2 placebo tablets). These doses are equivalent to 24/26 mg, 49/51 mg, and 97/103 mg commercial Entresto™, respectively. The doses of valsartan are 40mg (one 40 mg active and 1 placebo tablet), 80 mg (one 80 mg active and 1 placebo tablet), and 160 mg (two 80 mg active and 2 placebo tablets). The criteria for doubling the dose will be based on systolic blood pressure (a SBP > 90 mmHg is required for up titration), changes in renal function (maximum serum creatinine of 2.0 mg/dL), and the absence of symptoms of hypotension. For those not tolerating the current dose of study drug, the dose will be down-titrated to the previous tolerated dose. Subjects will return to clinic for follow-up visits at 2, 4, 8, 12, and 24 weeks after randomization.

Assessments at the follow-up visits include some or all of the following: interim medical history, review of medications, physical examination with the New York Heart Association (NYHA) class assessment, Kansas City Cardiomyopathy Questionnaire (KCCQ) quality of life questionnaire, local laboratory testing (creatinine, Blood Urea Nitrogen (BUN), electrolytes), Core laboratory testing (Cystatin C, BNP, NT-proBNP), adherence and tolerance assessment, and adverse event monitoring.

Follow-up phone calls will be made at 10, 16, and 20, weeks after randomization to assess dosing compliance, record the occurrence of applicable adverse events and events of interest, and remind the subject of the date and time of their next in-person visit.

A final phone visit is conducted approximately 2 weeks after study visit 10 (26 weeks after randomization) to assess clinical stability and any applicable adverse events.

During the consent process, subjects will be asked if interested in donating samples and data for research purposes via a biorepository and/or genetic study. Based on site and IRB preference, this optional part of the study may be incorporated into the main consent or may be a separate consent and Institutional Review Board (IRB) application.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced HFrEF defined as including ALL

   1. LVEF≤ 35% documented during the preceding 12 months
   2. NYHA class IV symptomatology, defined as chronic dyspnea or fatigue at rest or on minimal exertion in the previous 3 months, or patients who require chronic inotropic therapy
   3. Minimum of 3 months GDMT for HF and/or intolerant to therapy
2. Systolic blood pressure ≥ 90 mmHg
3. Serum NT-proBNP ≥ 800 pg/mL OR BNP ≥ 250 pg/mL (most recent - less than 3 months old)
4. Any one or more of the following objective findings of advanced HF including:

   1. Current inotropic therapy or use of inotropes in the past 6 months
   2. ≥ 1 hospitalization for heart failure in the past 6 months (not including the index hospitalization for inpatient participants)
   3. LVEF ≤ 25% (within the past 12 months)
   4. Peak VO2 < 55% predicted or peak VO2 ≤ 16 for men or ≤ 14 for women (Respiratory Exchange Ratio (RER) ≥ 1.05) (within the past 12 months)
   5. 6 min walk test distance < 300 m (within the past 3 months)
5. Age ≥18 years and ≤ 85 years
6. Signed Informed Consent form

Exclusion Criteria:

1. Currently taking Entresto™
2. History of hypersensitivity or intolerance (unmodifiable) to Entresto™, an ACEI or ARB as well as known or suspected contraindications (including hereditary angioedema) to the study drugs.
3. Estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73 m2 at baseline
4. Co-morbid conditions that may interfere with completing the study protocol (e.g. recent history of drug or alcohol abuse) or cause death within 1 year
5. Symptomatic hypotension at randomization or systolic blood pressure < 90 mmHg
6. Serum potassium > 5.5 mmol/L
7. Severe liver dysfunction (Childs-Pugh Class C)
8. Acute coronary syndrome within 4 weeks as defined by electrocardiographic (ECG) changes and biomarkers of myocardial necrosis (e.g. troponin) in an appropriate clinical setting (chest discomfort or anginal equivalent)
9. Planned or recent (≤ 4 weeks) PCI, coronary artery bypass grafting, or biventricular pacing
10. Currently hospitalized and listed status 1A, 1B or 1-4 for heart transplant
11. Current or scheduled for LVAD implantation within 30 days of study enrollment
12. Active infection (current use of oral or IV antimicrobial agents)
13. Primary hypertrophic or infiltrative cardiomyopathy, acute myocarditis, constrictive pericarditis or tamponade
14. Complex congenital heart disease
15. Concomitant use of aliskiren in patients with diabetes or renal impairment (eGFR <60 mL/min/1.73 m²)
16. Known pregnancy or anticipated pregnancy within the next 6 months or breastfeeding mothers
17. Enrollment in any other investigational clinical trial within 30 days prior to screening
18. Inability to comply with study procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Anstrom, Principal Investigator — Duke Health; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (38):
- United States (38):
  - Cedars-Sinai Heart Institute, Beverly Hills, California
  - Sutter Health Mills-Peninsula Health Services, Sacramento, California
  - San Diego Cardiac Center, San Diego, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Charlotte-Mecklenburg Hospital Authority, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Case Western Medical Center, Cleveland, Ohio
  - Metro Health System, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Geisinger Medical Center, Wilkes-Barre, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Research Institute, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Inova Heart and Vascular Insititute, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vader JM, Givertz MM, Starling RC, McNulty SE, Anstrom KJ, Desvigne-Nickens P, Hernandez AF, Braunwald E, Mann DL; LIFE Investigators. Tolerability of Sacubitril/Valsartan in Patients With Advanced Heart Failure: Analysis of the LIFE Trial Run-In. JACC Heart Fail. 2022 Jul;10(7):449-456. doi: 10.1016/j.jchf.2022.04.013. PMID 35772853
- [Derived] Mann DL, Givertz MM, Vader JM, Starling RC, Shah P, McNulty SE, Anstrom KJ, Margulies KB, Kiernan MS, Mahr C, Gupta D, Redfield MM, Lala A, Lewis GD, DeVore AD, Desvigne-Nickens P, Hernandez AF, Braunwald E; LIFE Investigators. Effect of Treatment With Sacubitril/Valsartan in Patients With Advanced Heart Failure and Reduced Ejection Fraction: A Randomized Clinical Trial. JAMA Cardiol. 2022 Jan 1;7(1):17-25. doi: 10.1001/jamacardio.2021.4567. PMID 34730769
- [Derived] Mann DL, Greene SJ, Givertz MM, Vader JM, Starling RC, Ambrosy AP, Shah P, McNulty SE, Mahr C, Gupta D, Redfield MM, Lala A, Lewis GD, Mohammed SF, Gilotra NA, DeVore AD, Gorodeski EZ, Desvigne-Nickens P, Hernandez AF, Braunwald E; LIFE Investigators. Sacubitril/Valsartan in Advanced Heart Failure With Reduced Ejection Fraction: Rationale and Design of the LIFE Trial. JACC Heart Fail. 2020 Oct;8(10):789-799. doi: 10.1016/j.jchf.2020.05.005. Epub 2020 Jun 10. PMID 32641226

RESULTS

PARTICIPANT FLOW:
Groups:
- LCZ696 (Entresto) + Placebo: LCZ696 50 mg, 100 mg, or 200 mg orally twice daily for 24 weeks, plus valsartan placebo (to match 40 mg, 80 mg, or 160 mg) orally twice daily for 24 weeks
  LCZ696: Subjects previously taking no or low-dose ACEI or ARB, or who have an eGFR < 30 mL/min/1.73m²: starting dose of LCZ696 = 50 mg po BID.
  Subjects taking an ARB at greater than low dose: starting dose of LCZ696 = 100 mg po BID.
  Subjects taking an ACEI at greater than low dose: starting dose of LCZ696 = 100 mg po BID.
  * At Investigator discretion, study drug may be started at the low dose if there are any concerns regarding tolerability.
  Dose adjustments will be performed every 2 weeks by doubling the dose of LCZ696 up to the target max dose of 200 mg po BID as tolerated.
  The doses of LCZ696 are 50mg (one low-dose (50mg) tablet), 100mg (one high-dose (100mg) tablet), and 200mg (two high-dose (100mg) tablets.) These doses are equivalent to 24/26 mg, 49/51 mg, and 97/103 mg commercial Entresto™, respectively.
  valsartan placebo: Valsartan placebo tablets will be supplied to match the low-dose (40mg) and high-dose (80mg) active valsartan tablets. Dosing for valsartan placebo will mirror dosing for active LCZ696 (the same number of low or high-dose tablets will be given.)
- Valsartan + Placebo: valsartan 40 mg, 80 mg, or 160 mg orally twice daily for 24 weeks, plus LCZ696 placebo (to match 50 mg, 100 mg, or 200 mg) orally twice daily for 24 weeks
  valsartan: Subjects previously taking no or low-dose ACEI or ARB, or who have an eGFR < 30 mL/min/1.73m²: the starting dose of valsartan = 40 mg po BID.
  Subjects taking an ARB at greater than low dose: starting dose of valsartan = 80 mg po BID.
  Subjects taking an ACEI at greater than low dose: starting dose of valsartan = 80 mg po BID.
  * At Investigator discretion, study drug may be started at the low dose if there are any concerns regarding tolerability.
  Dose adjustments will be performed every 2 weeks by doubling the dose of valsartan up to the target maximum dose of 160 mg po BID, as tolerated.
  The doses of valsartan are 40mg (one low-dose (40mg) tablet), 80mg (one high-dose (80mg) tablet), and 160mg (two high-dose (80mg) tablets).
  LCZ696 placebo: LCZ696 placebo tablets will be supplied to match the low-dose (50mg) and high-dose (100mg) active LCZ696 tablets. Dosing for LCZ696 placebo will mirror dosing for active valsartan (the same number of low or high-dose tablets will be given.)
Period: Overall Study
Arm/Group | LCZ696 (Entresto) + Placebo | Valsartan + Placebo
Started (Started is defined as randomized) | 179 | 186
Completed (Completed is defined as all patients that died or completed follow-up.) | 164 | 166
Not Completed | 15 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 (Entresto) + Placebo | Valsartan + Placebo | Total
Number analyzed (Participants) | 179 | 186 | 365
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (13.7) | 58.8 (13.0) | 59.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 50 | 103
  Male | 126 | 136 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 13 | 20
  Not Hispanic or Latino | 172 | 173 | 345
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 67 | 68 | 135
  White | 107 | 115 | 222
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 179 | 186 | 365

OUTCOME MEASURES:

1. Primary Outcome: Change in NT-proBNP
Description: The proportional change from baseline in the AUC for NT-proBNP levels measured at 2, 4, 8, 12, and 24 weeks. AUC was normalized for time and divided by the baseline value of NTproBNP so it has no unitshas no units. With the log-scale, the value of 0 indicates, on average, no change in NTproBNP from baseline. A value > 0 indicates an increase in log NT Pro BNP relative to baseline and a value < 0 indicates a decrease in log NT Pro BNP relative to baseline.
Time Frame: Baseline, 2, 4, 8, 12, and 24 weeks
Population: All randomized patients with baseline and at least one post-baseline NTpro BNP value present were included. Population was further reduced due to impact of COVID-19 by removing patients with inadequate follow-up after Feb 29th, 2020.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | LCZ696 (Entresto) + Placebo | Valsartan + Placebo
Number analyzed (Participants) | 155 | 158
unitless | 0.14 (0.65) | 0.19 (0.50)
Statistical Analysis 1: Comparison: LCZ696 (Entresto) + Placebo vs Valsartan + Placebo; AUC was normalized for time; With the log-scale, the value of 0 indicates, on average, no change in NTproBNP from baseline; Test type: Superiority; p = 0.45, Regression, Linear; ratio of the AUCs = 0.95, 95% CI 2-sided [0.84 to 1.08]

2. Secondary Outcome: Composite Endpoint of the Effects of LCZ696 (Number of Days)
Description: Composite endpoint of effects of LCZ696 compared to valsartan over 24 weeks will be compared based upon the number of days subjects are
  * alive and out of hospital
  * not listed for transplant (Status 1A, 1B or 1-4), or undergoing transplant
  * not implanted with an LVAD
  * not maintained or started on continuous inotropic therapy for ≥ 7 days
  * not hospitalized twice for HF (following the index admission) The days alive and out of hospital will end on the day of the second HF readmission, if applicable.
Time Frame: Randomization through 24 weeks
Population: Population was reduced due to impact of COVID-19 by removing patients with inadequate follow-up after Feb 29th, 2020.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | LCZ696 (Entresto) + Placebo | Valsartan + Placebo
Number analyzed (Participants) | 167 | 168
days | 108.58 [95.22 to 121.95] | 119.8 [107.64 to 131.96]
Statistical Analysis 1: Comparison: LCZ696 (Entresto) + Placebo vs Valsartan + Placebo; Test type: Superiority; p = 0.15, general linear model; Mean Difference (Net) = -11.22, 95% CI 2-sided [-26.4 to 3.97]

3. Secondary Outcome: Tolerability - Target Dose
Description: Tolerability as measured by number of subjects achieving a target dose of 0% (stopped study drug early or was never started on study drug), 25%, 50% or 100% of valsartan or LCZ696 (based on last dose of study drug taken prior to end of study)
Time Frame: Randomization through 24 weeks
Population: Population was reduced due to impact of COVID-19 by removing patients with inadequate follow-up after Feb 29th, 2020.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Entresto) + Placebo | Valsartan + Placebo
Number analyzed (Participants) | 167 | 168
Participants
  Not on study drug (0%) | 49 | 37
  Low dose (25%) | 28 | 41
  Mid dose (50%) | 33 | 30
  High dose (100%) | 57 | 60
Statistical Analysis 1: Comparison: LCZ696 (Entresto) + Placebo vs Valsartan + Placebo; Test type: Superiority; p = 0.51, ordinal logistic regression; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.78 to 1.68]

4. Secondary Outcome: Tolerability - Hypotension
Description: Tolerability as measured by number of subjects developing hypotension (SBP ≤ 85 mmHg) with symptoms
Time Frame: Randomization through 24 weeks
Population: Population was reduced due to impact of COVID-19 by removing patients with inadequate follow-up after Feb 29th, 2020.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Entresto) + Placebo | Valsartan + Placebo
Number analyzed (Participants) | 167 | 168
Participants
  Yes | 29 | 20
  No | 138 | 148
Statistical Analysis 1: Comparison: LCZ696 (Entresto) + Placebo vs Valsartan + Placebo; Test type: Superiority; p = 0.16, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.84 to 2.87]

5. Secondary Outcome: Tolerability - Renal Function
Description: Tolerability as measured by number of subjects developing worsening renal function (eGFR < 20 ml/min/1.73 m²)
Time Frame: Randomization through 24 weeks
Population: Population was reduced due to impact of COVID-19 by removing patients with inadequate follow-up after Feb 29th, 2020.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Entresto) + Placebo | Valsartan + Placebo
Number analyzed (Participants) | 167 | 168
Participants
  Yes | 7 | 7
  No | 160 | 161
Statistical Analysis 1: Comparison: LCZ696 (Entresto) + Placebo vs Valsartan + Placebo; Test type: Superiority; p = 0.99, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.34 to 2.91]

6. Secondary Outcome: Tolerability - Hyperkalemia
Description: Tolerability as measured by number of subjects developing moderate (>/= 5.5 mmol/L-5.9 mmol/L) or severe (>/= 6 mmol/L) hyperkalemia
Time Frame: Randomization through 24 weeks
Population: Population was reduced due to impact of COVID-19 by removing patients with inadequate follow-up after Feb 29th, 2020.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Entresto) + Placebo | Valsartan + Placebo
Number analyzed (Participants) | 167 | 168
Participants
  Yes | 28 | 15
  No | 139 | 153
Statistical Analysis 1: Comparison: LCZ696 (Entresto) + Placebo vs Valsartan + Placebo; Test type: Superiority; p = 0.035, Regression, Logistic; Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.05 to 4.00]

7. Other Pre Specified Outcome: Time to Death
Description: Time to death through 24 weeks
Time Frame: Randomization through 24 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Time to First Heart Failure (HF) Hospitalization
Description: Time to first HF hospitalization through 24 weeks
Time Frame: Randomization through 24 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Time to Death and First Heart Failure (HF) Hospitalization
Description: Time to death and first HF hospitalization through 24 weeks
Time Frame: Randomization through 24 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Total Number of Heart Failure (HF) Hospitalizations
Description: Total number of HF hospitalization admissions through 24 weeks
Time Frame: Randomization through 24 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Inotropic Therapy
Description: Number of subjects on continuous inotropic therapy >/= 7 days after discharge from the index hospitalization through 24 weeks
Time Frame: Randomization through 24 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Number of Subjects Listed for Transplant (Status 1A, 1B or 1-4), Transplanted or Implanted With an LVAD
Description: Number of subjects listed for transplant (status 1A, 1B or 1-4), transplanted or implanted with an LVAD through 24 weeks.
Time Frame: Randomization through 24 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in eGFR and Cystatin C Levels
Description: Change in eGFR and cystatin C levels compared to baseline. Renal function will be assessed at baseline, 4, 8, 12, and 24 weeks
Time Frame: Randomization through 24 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Unanticipated IV Diuretic Use
Description: Number of subjects with unanticipated use of IV diuretics (outpatient, ER or inpatient) through 24 weeks.
Time Frame: Randomization through 24 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in AUC in the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Difference in AUC of the KCCQ at 4, 12 and 24 weeks
Time Frame: Randomization through 24 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in AUC for the Ratio of NT-proBNP/BNP
Description: The change in AUC for the ratio of NT-proBNP/BNP from baseline to weeks 2, 4, 8, 12 and 24 weeks
Time Frame: Randomization through 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Randomization to week 24
Description: Adverse event collection was limited to those meeting serious criteria; SAEs were assessed at each study visit/phone call conducted. Population was reduced due to impact of COVID-19 by removing patients with inadequate follow-up after Feb 29th, 2020.
Arm/Group | LCZ696 (Entresto) + Placebo | Valsartan + Placebo
All-Cause Mortality (participants affected / at risk) | 13/167 | 8/168
Serious Adverse Events (participants affected / at risk) | 43/167 | 27/168
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCZ696 (Entresto) + Placebo (N=167) | Valsartan + Placebo (N=168)
Urinary Tract Obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal Haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Complication Associated With Device (General disorders) | 0 (0) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 4 (4) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Heart Transplant Rejection (Immune system disorders) | 0 (0) | 1 (1)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (2)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Arthritis Infective (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Infuenza (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3)
Pneumonia Klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Upper Respirator Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body In Gastrointestinal Tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anticoagulation Drug Level Below Therapeutic (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Device Dislocation (Product Issues) | 1 (1) | 0 (0)
Lead Dislodgement (Product Issues) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Substance Abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-Induced Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT02816736/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT02816736/SAP_001.pdf
  • Informed Consent Form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT02816736/ICF_002.pdf